CLINICAL TRIAL: NCT02724878
Title: Phase II Study of Atezolizumab + Bevacizumab in Patients With Advanced Non-Clear Cell Renal Cell Carcinoma
Brief Title: Study of Atezolizumab + Bevacizumab in Patients With Advanced Non-Clear Cell Renal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Toni Choueiri, MD, Toni K. Choueiri, MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-592
Record Dates: First submitted 2016-03-16; First posted 2016-03-31 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-01

CONDITIONS: Advanced Non-Clear Cell Kidney Cancer
Keywords: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Bevacizumab; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab And Atezolizumab Combination (Experimental): 1200 mg of Atezolizumab intravenously x 3 weeks
  15 mg/kg of Bevacizumab intravenously x 3 weeks.
  One cycle will be 3 weeks in duration.
  Interventions: Drug: Bevacizumab; Drug: Atezolizumab

INTERVENTIONS:
Drug: Bevacizumab
  Other Names: Avastin
Drug: Atezolizumab
  Other Names: RG-7446

SUMMARY:
This research study is studying the combination of Atezolizumab and Bevacizumab as a possible treatment for Advanced Non-Clear Cell Kidney Cancer.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. In this research the investigators are studying the combination of Atezolizumab with Bevacizumab. Participants will receive both vascular endothelial targeted therapy and immunotherapy.

The FDA (the U.S. Food and Drug Administration) has not approved Atezolizumab for Advanced Non-Clear Cell Kidney Cancer, but it has been approved for other uses.

The FDA has approved Bevacizumab with Interferon (IFNα) as a treatment option for Advanced Kidney Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Unresectable advanced or metastatic non-clear cell RCC to include but not limited to:

  * Papillary RCC, any type
  * Unclassified RCC
  * Translocation RCC
  * Chromophobe RCC
  * Collecting duct RCC
  * Medulary RCC
  * Clear cell RCC or any histology with > 20% sarcomatoid features will be eligible.
  * Other non-clear cell histologies that are not included above need to be discussed with the PI.
* Request for formalin-fixed, paraffin-embedded (FFPE) archival tumor specimens if available and willingness of the participant to undergo mandatory fresh tumor biopsy unless determined medically unsafe or not feasible. A note from the study team should be provided documenting availability of tissue. If a target lesion is biopsied at screening, this lesion must be followed as non-target lesion after the biopsy unless it is the patient's only target lesion. If there is only one target lesion, it should be followed as a target lesion regardless.

  * The archival specimen should contain adequate viable tumor tissue.
  * The specimen may consist of a tissue block (preferred and should contain the highest grade of tumor) or at least 30 unstained serial sections. Fine-needle aspiration, brushings, cell pellet from pleural effusion, bone marrow aspirate/biopsy are not acceptable.
  * Fresh tumor biopsy at progression will be required in cases where patients experience relapse after an initial response if medically safe.
* Measurable disease as defined by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
* ECOG performance status ≤ 2 (See Appendix A).
* Adequate hematologic and end-organ function as defined by the following laboratory results obtained within 28 days prior to the first study treatment:

  * Absolute neutrophil count (ANC) ≥ 1500 cells/uL.
  * Lymphocyte count ≥ 500/uL.
  * Platelet count ≥ 100,000/uL.
  * Hemoglobin ≥ 9 g/dL (patients may be transfused to meet this criterion).
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN) with the following exceptions: Patients with documented liver metastases should have AST and ALT ≤ 5 x ULN.
  * Serum bilirubin ≤ 2.0 x ULN with the following exception: Patients with known Gilbert's disease should have a serum bilirubin ≤ 3 x ULN.
  * Creatinine clearance ≥ 30 mL/min as calculated by Cockcroft-Gault equation.
* For female patients of childbearing potential and male patients with partners of childbearing potential, agreement (by patient and/or partner) to use highly effective forms of contraception and to continue its use 6 months after the last dose of atezolizumab or bevacizumab.
* Signed informed consent form.
* Ability and capacity to comply with study and follow-up procedures.

Exclusion Criteria

•Prior treatment with CD137 agonists, anti- cytotoxic T-lymphocyte-associated protein 4, anti-PD-1, or anti-PDL1 therapeutic antibody or pathway targeting agents.

Prior IFNα or IL-2 is allowed following 4 week washout from treatment end date.

* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitors) within 2 weeks of enrollment or receipt of any anti-cancer therapy (including investigational therapy, monoclonal antibodies, cytokine therapy) within 4 weeks of enrollment.
* Prior therapy with bevacizuamab.
* Thrombologic event within 3 weeks of treatment start date, unless stable on anticoagulation with LMWH or Factor Xa inhibitor for at least 2 weeks.
* Treatment with systemic immunosuppressive medications including but not limited to: prednisone, dexamethasone, cyclosporin, azathioprine, methotrexate, thalidomide, anti- tumor necrosis factor (TNF) agents, hydroxychloroquine within 2 weeks of first study dose.

  * Patients who have received acute, low-dose systemic immunosuppressant medications may be enrolled.
  * Patients with adrenal insufficiency on physiologic replacement doses of steroids may be enrolled.
  * The use of inhaled, topical intraocular, or intra articular corticosteroids or, mineralocorticoids are allowed.
* Radiotherapy for RCC within 14 days of first study treatment with the exception of a single fraction of radiation administered for palliation of symptoms.
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy, radiosurgery, or surgery and stable for at least 4 weeks prior to the initiation of study treatment. Stability must be confirmed by magnetic resonance imaging (MRI) or computed tomography (CT) imaging and/or treating investigator determination.
* Malignancies other than RCC within 2 years of first study treatment with the exception of those with negligible risk of metastases or death (included but not limited to carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, ductal carcinoma in situ of the breast, non-muscle invasive urothelial carcinoma, or other malignancy not deemed to impact that patients 5-year life expectancy).
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion protein.
* Known hypersensitivity to any component of the atezolizumab product.
* History of autoimmune disease including: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, Wegner's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, type I diabetes mellitus, vasculitis, or glomerulonephritis. Patients with a history of autoimmune-related hypothyroidism on thyroid replacement hormone or those with autoimmune dermatologic conditions not requiring the use of prednisone > 10 mg or equivalent are eligible.
* History of idiopathic pulmonary fibrosis, organized pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening imaging CT of the chest. History of radiation pneumonitis in the radiation field is permitted.
* Positive test for HIV (test to be performed within 28 days of first treatment start).
* Patients with active or chronic hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening). Patients with past/resolved HBV infection (defined as having negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible. A negative HBA DNA test must be obtained in patients with positive hepatitis B core antibody prior to Cycle 1 Day 1.
* Active hepatitis C infection. Patients positive hepatitis C antibody test are eligible if PCR is negative for hepatitis C viral DNA.
* Infection requiring receipt of therapeutic oral or IV anti-microbials within 2 weeks of first study treatment. Patients receiving routine anti-microbial prophylaxis (for dental extractions/procedures) are eligible.
* Significant cardiovascular disease such as New York Heart Association (NYHA) class II or greater, myocardial infarction within the previous 3 months of first study treatment, unstable arrhythmias, unstable angina. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 50% must be on a stable regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist when appropriate.
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg). Anti-hypertensive therapy to achieve these parameters is allowed.
* Prior history of hypertensive crisis or hypertensive encephalopathy within the previous 3 months of first study treatment.
* History of stroke or transient ischemic attack within 3 months of first study dose.
* Significant vascular disease (such as aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months of first study dose. Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* Current or recent use of dipyramidole, ticlopidine, clopidogrel, cilostazol is excluded. Aspirin (≤ 325 mg per day) is allowed. Prophylactic anticoagulation with oral or parenteral anticoagulants for the patency of venous access devices or other indications is allowed. Therapeutic use of low-molecular weight heparin (such as enoxaparin), and factor Xa inhibitors are allowed. Use of warfarin is prohibited.
* Use of plaquenil must be discontinued two weeks prior to first study treatment.
* History of abdominal or tracheoesophageal fistula or GI perforation within 6 months of first study treatment.
* Clinical signs or symptoms of active GI obstruction or requirement of routine parenteral nutrition or tube feedings.
* Evidence of abdominal free air not explained by paracentesis or recent surgical procedure.
* Serious, non-healing or dehiscing wound or active ulcer.
* Proteinuria, as demonstrated by > 1.5 gram of protein in a 24-hour urine collection. All patients with ≥ 2+ protein on dipstick urinalysis at baseline must undergo 24-hour urine collection for protein.
* Major surgical procedure within 21 days of first study treatment.
* Prior allogenic stem cell or solid organ transplant.
* Administration of a live, attenuated vaccine within 4 weeks for first study treatment.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toni Choueiri, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - University of California, San Diego Moores Cancer Center, La Jolla, California
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Available upon request.

REFERENCES:
- [Background] Saliby RM, El Zarif T, Bakouny Z, Shah V, Xie W, Flippot R, Denize T, Kane MH, Madsen KN, Ficial M, Hirsch L, Wei XX, Steinharter JA, Harshman LC, Vaishampayan UN, Severgnini M, McDermott DF, Lee GM, Xu W, Van Allen EM, McGregor BA, Signoretti S, Choueiri TK, McKay RR, Braun DA. Circulating and Intratumoral Immune Determinants of Response to Atezolizumab plus Bevacizumab in Patients with Variant Histology or Sarcomatoid Renal Cell Carcinoma. Cancer Immunol Res. 2023 Aug 3;11(8):1114-1124. doi: 10.1158/2326-6066.CIR-22-0996. PMID 37279009
- [Result] McGregor BA, McKay RR, Braun DA, Werner L, Gray K, Flaifel A, Signoretti S, Hirsch MS, Steinharter JA, Bakouny Z, Flippot R, Wei XX, Choudhury A, Kilbridge K, Freeman GJ, Van Allen EM, Harshman LC, McDermott DF, Vaishampayan U, Choueiri TK. Results of a Multicenter Phase II Study of Atezolizumab and Bevacizumab for Patients With Metastatic Renal Cell Carcinoma With Variant Histology and/or Sarcomatoid Features. J Clin Oncol. 2020 Jan 1;38(1):63-70. doi: 10.1200/JCO.19.01882. Epub 2019 Nov 13. PMID 31721643

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place between July 2016 and October 2018.
Period: Overall Study
Arm/Group | Bevacizumab And Atezolizumab Combination
Started | 65
Treated | 60
Responders | 20
Completed | 0
Not Completed | 65
Not completed — Still on Active Therapy | 15
Not completed — Disease Progression | 31
Not completed — Toxicity | 5
Not completed — Death | 1
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 2
Not completed — Protocol Violation | 1
Not completed — Ineligible for Study Drug | 5
Not completed — not started | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
Age, Continuous [Median (Full Range); unit: years] | 61 [22 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 56
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 53
  More than one race | 2
  Unknown or Not Reported | 2
Metastasis Stage at Diagnosis [Number; unit: participants] — Stages:
  * M0: Cancer has not spread to other parts of the body.
  * M1: Cancer has spread to other parts of the body.
  participants
    M0 | 8
    M1 | 16
    Unknown | 36
Histology [Count of Participants; unit: Participants]
  Clear Cell | 18
  Papillary | 12
  Chromophobe | 10
  Unclassified | 9
  Transcription Factor E3 Translocation | 5
  Collecting Duct | 5
  Medullary | 1
Sarcomatoid Differentiation [Count of Participants; unit: Participants] | 26
ECOG Performance Status [Count of Participants; unit: Participants]
  00 - Fully Active | 29
  01 - Restricted | 30
  02 - Ambulatory and Capable of Self Care | 1
Prior Nephrectomy [Count of Participants; unit: Participants] | 52
Prior Systemic Therapy [Count of Participants; unit: Participants] | 21
Presence of Bone Metastases [Count of Participants; unit: Participants] | 1
Presence of Liver Metastases [Count of Participants; unit: Participants] | 11
International Metastatic Renal Cell Carcinoma Database Consortium Risk Group [Count of Participants; unit: Participants]
  Favorable | 9
  Intermediate | 33
  Poor | 18

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate
Description: The best overall response rate is the percentage of participants achieving complete response (CR) or partial response (PR) as the best response recorded on treatment based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria.
  CR and PR must meet the following lesion criteria without having any new lesions as well:
  Target Lesion:
  (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
  Non-Target Lesion:
  (CR): Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).
  Non-CR/Non-Progressive Disease: Persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. Must have PR in target lesion.
Time Frame: Measured every 6 weeks for the first 24 weeks and then every 12 weeks while on treatment. The median (range) of treatment time was 9.5 (1-42) cycles, thus participants were assessed up to ~32 months .
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
percentage of participants | 33 [25 to 42]
Statistical Analysis 1: Comparison: Bevacizumab And Atezolizumab Combination; A sample size of 60 would provide 95% power to distinguish the ORR rate of 25% from 10% (historical control) with 1-sided alpha of 0.07. The treatment would be considered effective if 10 or more responses are observed out of 60 patients; Test type: Superiority; Response Rate = 33, 80% CI 2-sided [25 to 42]

2. Secondary Outcome: Best Overall Response Rate by Histological Subtypes
Description: The best overall response rate is the percentage of participants achieving complete response (CR) or partial response (PR) as the best response recorded on treatment based on Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria. Please see the primary endpoint "Best Overall Response Rate" description for the definition of CR and PR.
  Non-clear cell renal cell carcinoma includes different histologic and genetic subtypes to include: papillary, chromophobe, collecting duct, unclassified, translocation, and medullary carcinoma. These subtypes are measured using established methods.
Time Frame: Measured every 6 weeks for the first 24 weeks and then every 12 weeks while on treatment. The median (range) of treatment time was 9.5 (1-42) cycles, thus participants were assessed up to ~32 months
Population: The number analyzed for each row is less than 60 because each row represents a histological subgroup. The sum of number analyzed by row equals the total number analyze (60).
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
percentage of participants
  Papillary: number analyzed (Participants) | 12
  Papillary | 23 [10 to 48]
  Chromophobe: number analyzed (Participants) | 10
  Chromophobe | 10 [1 to 34]
  Unclassified: number analyzed (Participants) | 9
  Unclassified | 33 [13 to 60]
  Transcription Factor E3 Translocation: number analyzed (Participants) | 5
  Transcription Factor E3 Translocation | 20 [2 to 58]
  Collecting Duct: number analyzed (Participants) | 5
  Collecting Duct | 40 [12 to 77]
  Medullary: number analyzed (Participants) | 1
  Medullary | 100 [10 to 100]
  Clear Cell: number analyzed (Participants) | 18
  Clear Cell | 50 [33 to 67]

3. Secondary Outcome: Percentage of Participants With Treatment-related Adverse Events
Description: Assessed by -Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. All treatment-related all-grade adverse events occurring in >10% of participants.
  Treatment Related is discerned as follows:
  * Yes: There is a plausible temporal relationship between the onset of the AE and administration of atezolizumab or bevacizumab, and the AE cannot be readily explained by the patient's clinical state, intercurrent illness, or concomitant therapies; and/or the AE follows a known pattern of response to atezolizumab or bevacizumab or with similar treatments; and/or the AE resolves upon discontinuation of the study drugs or dose reduction and, if applicable, reappears upon re-challenge.
  * No: Evidence exists that the AE has an etiology other than the study drugs (e.g., pre existing medical condition, underlying disease, intercurrent illness, or concomitant medication); and/or the AE has no plausible temporal relationship to the study drugs administration.
Time Frame: Adverse events are measured continuously on treatment and up to thirty days after going off treatment (up to ~32 months).
Population: The analysis population is comprised of all treated patients.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
percentage of participants
  Fatigue | 35
  Proteinuria | 35
  Musculoskeletal Pain | 33
  Diarrhea | 22
  Rash | 20
  Hypertension | 18
  Pruritis | 18
  Thyroid Dysfunction | 17
  Hepatitis | 15
  Fever | 13
  Mucositis | 12

4. Secondary Outcome: Duration of Response
Description: The duration of overall response (based on RECIST 1.1) is measured from the time measurement criteria are met for CR and PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented taking as reference for progressive disease the smallest measurements recorded since the treatment started or death due to any cause. Participants without events reported are censored at the last disease evaluation.
Time Frame: Measured every 6 weeks for the first 24 weeks and then every 12 weeks while on treatment. Off-treatment, patients are followed every 6 months for up to two year. Participants were followed up to 32 months.
Measure: Median (Full Range); unit: months
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 20
months | 8.9 [1.4 to 29]

5. Secondary Outcome: Immune Related Best Overall Response Rate
Description: The best overall Immune-Related Complete Response (irCR) or Immune-Related Partial Response (irPR) is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
  irCR: Complete disappearance of all target lesions in two consecutive observations not less than 4 weeks apart. This category encompasses exactly the same subjects as complete response (CR).
  irPR: Decrease, relative to baseline, of 50% or greater in the sum of the products of the two largest perpendicular diameters (SPD) of all target and all new measurable lesions in two consecutive observations not less than 4 weeks apart. Note: the appearance of new measurable lesions is factored into the overall tumor burden, but does not automatically qualify as progressive disease until the SPD increases by > 25% when compared to SPD at nadir.
Time Frame: Measured every 6 weeks while on treatment. Off-treatment, patients are followed every 6 months for up to two year. Participants were followed up to 32 months.
Population: Since the trial was designed in 2015, immune-related response has been infrequently used in VEGF/IO trials for kidney cancer. Most RCC trials have mainly focused on the traditional RECIST-based response as the primary endpoint. Therefore, the study team did not pursue immune-related response assessment and that data was not collected.
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 0

6. Secondary Outcome: Median Progression Free Survival
Description: Progression free survival (PFS) is defined as the time from start of treatment to disease progression (PD) or death from any cause as estimated by Kaplan Meier methods. Patients who have not progressed and are alive are censored at the date the patient is known to be progression-free. Progression is defined by Response Evaluation Criteria In Solid Tumors Criteria 1.1 (RECIST) as follows:
  - >20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (including baseline if it's the smallest). The sum must also demonstrate an increase of >5 mm.
  OR
  -Appearance of new lesions and/or unequivocal progression of non-target lesions. It must be representative of overall disease status change, not a single lesion increase. For patients with PD at the first on-treatment imaging assessment, patients will be allowed to remain on study until confirmation at the next assessment at investigator discretion if patient is benefiting from treatment.
Time Frame: Participants followed for up to 32 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
months | 8.3 [5.7 to 10.9]

7. Secondary Outcome: 1-Year Overall Survival
Description: 1-Year Overall Survival (OS) is defined as the probability of survival at 1 year from treatment start date. Survival probability is estimated using Kaplan Meier methods. An event is considered to be death due to any cause. Participants who are lost to follow-up before the 1 year mark are censored at date last known alive.
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percent probability of survival
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
percent probability of survival | 67 [52 to 79]

8. Secondary Outcome: Mean Function Assessment of Cancer Therapy-Kidney Symptom Index-19 Score
Description: The Function Assessment of Cancer Therapy-Kidney Symptom Index-19 (FKSI-19) is a 19 item questionnaire with each item scored on a scale of 0-4 for a total score of 0-76 with higher scores indicating fewer symptom.
Time Frame: Assessed at baseline, week 3, week 5, week 7, week 9, and end of therapy.
Population: Number analyzed reflects the number of participants with a evaluable questionnaire at each timepoint.
Measure: Mean (Inter-Quartile Range); unit: score on scale
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
score on scale
  Baseline | 55.72 [48.0 to 64.0]
  3 weeks: number analyzed (Participants) | 45
  3 weeks | 59.13 [54.0 to 65.0]
  5 weeks: number analyzed (Participants) | 40
  5 weeks | 59.13 [61.0 to 67.0]
  7 weeks: number analyzed (Participants) | 36
  7 weeks | 60.66 [52.0 to 70.0]
  9 weeks: number analyzed (Participants) | 33
  9 weeks | 62.41 [55.0 to 70.0]
  End of Therapy: number analyzed (Participants) | 29
  End of Therapy | 51.92 [44.0 to 59.0]

9. Secondary Outcome: Brief Fatigue Inventory Score - Items 1-3
Description: The Brief Fatigue Inventory Score (BFI) is a 9 item questionnaire with each items 1-3 scored on a scale of 0-10 Scores are categorized is mild (1-3), moderate (4-6), or severe (7-10). A global fatigue score can be found by averaging the score obtained on each test item completed. Items 1-3 of the 9 are reported here.
Time Frame: Assessed at baseline, week 9, week 15, week 21, week 27, and end of therapy.
Population: Number analyzed reflects the number of participants with a evaluable questionnaire at each timepoint. Items 1-3 are reported because they are fatigue related and fatigue is the most common toxicity in the cohort.
Measure: Mean (Inter-Quartile Range); unit: score on scale
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
score on scale
  Baseline: number analyzed (Participants) | 58
  Baseline | 3.56 [1.0 to 5.3]
  Week 9: number analyzed (Participants) | 42
  Week 9 | 3.44 [1.0 to 5.3]
  Week 15: number analyzed (Participants) | 38
  Week 15 | 3.25 [1.0 to 5.3]
  Week 21: number analyzed (Participants) | 34
  Week 21 | 2.97 [1.3 to 4.7]
  Week 27: number analyzed (Participants) | 30
  Week 27 | 2.70 [0.7 to 4.0]
  End of Therapy: number analyzed (Participants) | 13
  End of Therapy | 3.97 [3.0 to 6.0]

10. Secondary Outcome: 6-Month Progression-Free Survival by Histological Subgroups
Description: 6-Month Progression free survival (PFS) is defined as the probability of disease progression (PD) or death from any cause 6 months from treatment start date as estimated by Kaplan Meier methods. Patients who have not progressed and alive are censored at the date the patient is known to be progression-free. Progression is defined by RECIST 1.1 as follows:
  - >20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The sum must also demonstrate an increase of >5 mm.
  OR
  -Appearance of new lesions and/or unequivocal progression of non-target lesions. It must be representative of overall disease status change, not a single lesion increase. For patients with PD at the first on-treatment imaging assessment, patients will be allowed to remain on study until confirmation at the next assessment at investigator discretion if patient is benefiting from treatment.
  Histological subgroups are categorized using established methods.
Time Frame: 6 months
Population: Each row represent a histological subgroup
Measure: Number (95% Confidence Interval); unit: percent probability of PFS
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
percent probability of PFS
  Clear Cell: number analyzed (Participants) | 18
  Clear Cell | 58 [31 to 77]
  Papillary: number analyzed (Participants) | 12
  Papillary | 75 [41 to 91]
  Other clear cell Renal Cell Carcinoma: number analyzed (Participants) | 30
  Other clear cell Renal Cell Carcinoma | 59 [39 to 74]

11. Secondary Outcome: 1-Year Overall Survival by Histological Subgroup
Description: as for outcome 7
Time Frame: 1 year
Population: Each row represents a Histology subgroup.
Measure: Number (95% Confidence Interval); unit: percent probability of survival
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
percent probability of survival
  Clear Cell: number analyzed (Participants) | 18
  Clear Cell | 63 [35 to 82]
  Papillary: number analyzed (Participants) | 12
  Papillary | 79 [36 to 94]
  Other non-clear cell Renal Cell Carcinoma: number analyzed (Participants) | 30
  Other non-clear cell Renal Cell Carcinoma | 68 [46 to 82]

12. Secondary Outcome: 6-Month Progression-Free Survival by Sarcomatoid Differentiation
Description: 6-Month Progression free survival (PFS) is defined as the probability of disease progression (PD) or death from any cause 6 months from treatment start date as estimated by Kaplan Meier methods. Patients who have not progressed and alive are censored at the date the patient is known to be progression-free. Progression is defined by RECIST 1.1 as follows:
  - >20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The sum must also demonstrate an increase of >5 mm.
  OR
  -Appearance of new lesions and/or unequivocal progression of non-target lesions. It must be representative of overall disease status change, not a single lesion increase. For patients with PD at the first on-treatment imaging assessment, patients will be allowed to remain on study until confirmation at the next assessment at investigator discretion if patient is benefiting from treatment.
  Sarcomatoid Differentiation are categorized using established methods
Time Frame: 6 months
Population: Each row represents a Sarcomatoid Differentiation category.
Measure: Number (95% Confidence Interval); unit: percent probability of PFS
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
percent probability of PFS
  Sarcomatoid in clear cell Renal Cell Carcinoma: number analyzed (Participants) | 18
  Sarcomatoid in clear cell Renal Cell Carcinoma | 58 [31 to 77]
  Sarcomatoid in non-clear cell Renal Cell Carcinoma: number analyzed (Participants) | 8
  Sarcomatoid in non-clear cell Renal Cell Carcinoma | 38 [9 to 67]
  None: number analyzed (Participants) | 34
  None | 70 [51 to 82]

13. Secondary Outcome: 1-Year Overall Survival by Sarcomatoid Differentiation
Description: as for outcome 7
Time Frame: 1 year
Population: Each row represents a Sarcomatoid Differentiation category.
Measure: Number (95% Confidence Interval); unit: percent probability of survival
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
percent probability of survival
  Sarcomatoid in clear cell Renal Cell Carcinoma: number analyzed (Participants) | 18
  Sarcomatoid in clear cell Renal Cell Carcinoma | 63 [35 to 82]
  Sarcomatoid in non-clear cell Renal Cell Carcinoma: number analyzed (Participants) | 8
  Sarcomatoid in non-clear cell Renal Cell Carcinoma | 36 [1 to 78]
  None: number analyzed (Participants) | 34
  None | 74 [54 to 87]

14. Secondary Outcome: Objective Response Rate by Sarcomatoid Differentiation
Description: The objective response rate is the percentage of participants achieving complete response (CR) or partial response (PR) as the best response on treatment using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1).
  CR and PR must meet the following criteria without having any new lesions as well:
  Target Lesion:
  (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  (PR): >=30% decrease in the sum of the diameters of target lesion, taking as reference the baseline sum diameter.
  Non-Target Lesion:
  (CR): Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological (<10 mm short axis) Non-CR/Non-Progressive Disease: Persistence of 1+ non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. Must have PR in target lesion Sarcomatoid Differentiation are categorized using established methods
Time Frame: as for outcome 1
Population: Each row represents a Sarcomatoid Differentiation category.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
percentage of participants
  None: number analyzed (Participants) | 34
  None | 26 [17 to 36]
  Clear Cell Renal Carcinoma: number analyzed (Participants) | 18
  Clear Cell Renal Carcinoma | 50 [35 to 65]
  Variant Histology Renal Cell Carcinoma: number analyzed (Participants) | 8
  Variant Histology Renal Cell Carcinoma | 38 [16 to 60]

15. Secondary Outcome: 6-Month Progression-Free Survival by International Metastatic Renal Cell Carcinoma Risk Group
Description: 6-Month Progression free survival (PFS) is defined as the probability of disease progression (PD) or death from any cause 6 months from treatment start date as estimated by Kaplan Meier methods. Patients who have not progressed and alive are censored at the date the patient is known to be progression-free. Progression is defined by RECIST 1.1 as follows:
  - >20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum. The sum must also demonstrate an increase of >5 mm.
  OR
  -Appearance of new lesions and/or unequivocal progression of non-target lesions. It must be representative of overall disease status change, not a single lesion increase. For patients with PD at the first on-treatment imaging assessment, patients will be allowed to remain on study until confirmation at next assessment at investigator discretion if patient is benefiting from treatment.
  International Metastatic Renal Cell Carcinoma Risk Group determined by established methods
Time Frame: 6 months
Population: Each row represents an International Metastatic Renal Cell Carcinoma Risk Group
Measure: Number (95% Confidence Interval); unit: percent probability of PFS
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
percent probability of PFS
  Favorable: number analyzed (Participants) | 9
  Favorable | 78 [36 to 94]
  Intermediate: number analyzed (Participants) | 33
  Intermediate | 79 [61 to 89]
  Poor: number analyzed (Participants) | 18
  Poor | 19 [5 to 40]

16. Secondary Outcome: 1-Year Overall Survival by International Metastatic Renal Cell Carcinoma Risk Group
Description: as for outcome 7
Time Frame: 1 year
Population: Each row represents an International Metastatic Renal Cell Carcinoma Risk Group
Measure: Number (95% Confidence Interval); unit: percent probability of survival
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
percent probability of survival
  Favorable: number analyzed (Participants) | 9
  Favorable | 100 [100 to 100]
  Intermediate: number analyzed (Participants) | 33
  Intermediate | 79 [57 to 90]
  Poor: number analyzed (Participants) | 18
  Poor | 28 [8 to 53]

17. Secondary Outcome: Objective Response Rate by International Metastatic Renal Cell Carcinoma Risk Group
Description: The objective response rate is the percentage of participants achieving complete response (CR) or partial response (PR) as the best response on treatment using RECIST 1.1.
  CR and PR must meet the following criteria without having any new lesions as well:
  Target Lesion:
  (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  (PR): >=30% decrease in the sum of the diameters of target lesion, taking as reference the baseline sum diameter.
  Non-Target Lesion:
  (CR): Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological (<10 mm short axis).
  Non-CR/Non-Progressive Disease: Persistence of 1+ non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. Must have PR in target lesion.
  International Metastatic Renal Cell Carcinoma Risk Group are categorized using established methods
Time Frame: as for outcome 1
Population: Each row represents an International Metastatic Renal Cell Carcinoma Risk Group
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
percentage of participants
  Favorable: number analyzed (Participants) | 9
  Favorable | 33 [13 to 53]
  Intermediate: number analyzed (Participants) | 33
  Intermediate | 45 [35 to 57]
  Poor: number analyzed (Participants) | 18
  Poor | 11 [1.6 to 21]

18. Secondary Outcome: 6-Month Progression-Free Survival by Prior Systemic Therapy
Description: 6-Month Progression free survival (PFS) is defined as the probability of disease progression (PD) or death from any cause 6 months from treatment start date as estimated by Kaplan Meier methods. Patients who have not progressed and alive are censored at the date the patient is known to be progression-free. Progression is defined by RECIST 1.1 as follows:
  - >20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study. The sum must also demonstrate an increase of >5 mm.
  OR
  -Appearance of new lesions and/or unequivocal progression of non-target lesions. It must be representative of overall disease status change, not a single lesion increase. For patients with PD at the first on-treatment imaging assessment, patients will be allowed to remain on study until confirmation at the next assessment at investigator discretion if patient is benefiting from treatment.
  Prior systemic therapy group determined by established methods,
Time Frame: 6 months
Population: Each row represents a prior systemic therapy category.
Measure: Number (95% Confidence Interval); unit: percent probability of PFS
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
percent probability of PFS
  No: number analyzed (Participants) | 39
  No | 56 [39 to 71]
  Yes: number analyzed (Participants) | 21
  Yes | 71 [47 to 86]

19. Secondary Outcome: 1-Year Overall Survival by Prior Systemic Therapy
Description: as for outcome 7
Time Frame: 1 year
Population: Each row represents a prior systemic therapy category.
Measure: Number (95% Confidence Interval); unit: percent probability of survival
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
percent probability of survival
  No: number analyzed (Participants) | 39
  No | 66 [48 to 80]
  Yes: number analyzed (Participants) | 21
  Yes | 66 [33 to 85]

20. Secondary Outcome: Objective Response Rate by Prior Systemic Therapy
Description: The objective response rate is the percentage of participants achieving complete response (CR) or partial response (PR) as the best response on treatment using RECIST 1.1.
  CR and PR must meet the following criteria without having any new lesions as well:
  Target Lesion:
  (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  (PR): >=30% decrease in the sum of the diameters of target lesion, taking as reference the baseline sum diameter.
  Non-Target Lesion:
  (CR): Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological (<10 mm short axis).
  Non-CR/Non-Progressive Disease: Persistence of 1+ non-target lesion(s) and/or maintenance of tumor marker level above the normal limits. Must have PR in target lesion.
Time Frame: as for outcome 1
Population: Each row represents a prior systemic therapy category.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab And Atezolizumab Combination
Number analyzed (Participants) | 60
percentage of participants
  Yes: number analyzed (Participants) | 39
  Yes | 31 [25 to 52]
  No: number analyzed (Participants) | 21
  No | 38 [21 to 40]

ADVERSE EVENTS:
Time Frame: Adverse events are measured continuously on treatment and up to thirty days after going off treatment (up to ~32 months).
Description: An adverse event (AE) was classified as serious (SAE) if any of the following are true:
  * It results in death or is life threatening.
  * It requires or prolongs inpatient hospitalization.
  * It results in persistent or significant disability/incapacity .
  * It results in a congenital anomaly/birth defect in a neonate/infant born to a mother.
  exposed to the IMP.
  - It is considered a significant medical event by the investigator based on medical judgment.
Arm/Group | Bevacizumab And Atezolizumab Combination
All-Cause Mortality (participants affected / at risk) | 19/60
Serious Adverse Events (participants affected / at risk) | 5/65
Other Adverse Events (participants affected / at risk) | 62/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab And Atezolizumab Combination (N=65)
Alkaline phosphatase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Pericardial effusion (Cardiac disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Multi-organ failure (General disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Hip fracture (Injury, poisoning and procedural complications) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab And Atezolizumab Combination (N=65)
Anemia (Blood and lymphatic system disorders) | 16
Leukocytosis (Blood and lymphatic system disorders) | 2
Lymph node pain (Blood and lymphatic system disorders) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 4
Atrial fibrillation (Cardiac disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Vertigo (Ear and labyrinth disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 2
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 18
Endocrine disorders - Other, specify (Endocrine disorders) | 1
Blurred vision (Eye disorders) | 2
Cataract (Eye disorders) | 1
Floaters (Eye disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 12
Ascites (Gastrointestinal disorders) | 4
Bloating (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Colonic fistula (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 21
Diarrhea (Gastrointestinal disorders) | 26
Dry mouth (Gastrointestinal disorders) | 4
Duodenal ulcer (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 2
Gastroparesis (Gastrointestinal disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 3
Lip pain (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 24
Oral dysesthesia (Gastrointestinal disorders) | 1
Oral hemorrhage (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 2
Stomach pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 13
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 5
Chills (General disorders) | 2
Edema limbs (General disorders) | 9
Fatigue (General disorders) | 51
Fever (General disorders) | 12
Flu like symptoms (General disorders) | 4
Gait disturbance (General disorders) | 1
Infusion related reaction (General disorders) | 4
Localized edema (General disorders) | 5
Multi-organ failure (General disorders) | 1
Neck edema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 11
General disorders and administration site conditions - Other, specify (General disorders) | 5
Portal vein thrombosis (Hepatobiliary disorders) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Allergic reaction (Immune system disorders) | 1
Autoimmune disorder (Immune system disorders) | 1
Bronchial infection (Infections and infestations) | 2
Catheter related infection (Infections and infestations) | 1
Conjunctivitis infective (Infections and infestations) | 1
Gum infection (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 1
Rhinitis infective (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Skin infection (Infections and infestations) | 2
Upper respiratory infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 3
Hip fracture (Injury, poisoning and procedural complications) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 10
Alkaline phosphatase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 14
Blood bilirubin increased (Investigations) | 3
Cholesterol high (Investigations) | 2
Creatinine increased (Investigations) | 11
Lipase increased (Investigations) | 1
Lymphocyte count decreased (Investigations) | 2
Lymphocyte count increased (Investigations) | 1
Platelet count decreased (Investigations) | 3
Serum amylase increased (Investigations) | 1
Weight gain (Investigations) | 2
Weight loss (Investigations) | 8
Acidosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 15
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 12
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 34
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 8
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 5
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amnesia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 4
Dysphasia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 14
Memory impairment (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 4
Somnolence (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 9
Confusion (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 12
Acute kidney injury (Renal and urinary disorders) | 4
Chronic kidney disease (Renal and urinary disorders) | 5
Hematuria (Renal and urinary disorders) | 2
Proteinuria (Renal and urinary disorders) | 27
Urinary frequency (Renal and urinary disorders) | 6
Urinary tract obstruction (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Gynecomastia (Reproductive system and breast disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 18
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 24
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 4
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 4
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 13
Rash acneiform (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Skin atrophy (Skin and subcutaneous tissue disorders) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 7
Flushing (Vascular disorders) | 1
Hematoma (Vascular disorders) | 2
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 23
Hypotension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT02724878/Prot_SAP_000.pdf